CLINICAL TRIAL: NCT02226523
Title: The Development and Clinical Application of Rapid Assays Using Multi-antibody-activated Magnetic Nanoparticles System in Acute Coronary Syndrome
Brief Title: Magnetic Nanoparticles System in Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Yen-Wen Wu, Chief of Cardiology Division of Cardiovascular Medical Center and Department of Nuclear Medicine, Far Eastern Memorial Hospital
Other Study IDs: 103002_N_103CT1026
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Acute Coronary Syndrome
Keywords: immunomagnetic reduction; acute coronary syndrome; serum biomarkers
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — plasma/serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To improve the sensitivity and specificity of immunoassay, the developing trends are to lower the detection threshold and to minimize the cross reaction. A new assay technology called immunomagnetic reduction (IMR) has been developed for rapid and on-site assay with small volume of sample. Rapid diagnosis of acute coronary syndrome (ACS) is a clinical and operational priority in busy emergency departments (ED), early and correct diagnosis is important. Cardiac enzymes (including CPK/CK-MB, troponins, myoglobulin) and electrocardiography (ECG) in combination with the medical history and physical examination are at present the diagnostic cornerstones. Novel biomarkers that rise earlier, have good diagnosis accuracy and have additional prognostic information are highly needed. The combination of multiple biomarker assays (markers of myocardial injury, inflammation/plaque ruptures or heart failure with different mechanism) may increase clinical sensitivity and improve early risk stratification. The present study, a rapid IMR assay with multiple biomarkers is proposed and we will examine the performance of this new investigational IMR assays, comparison with current commercial assays.

DETAILED DESCRIPTION:
To improve the sensitivity and specificity of immunoassay, the developing trends are to lower the detection threshold and to minimize the cross reaction. A new assay technology called immunomagnetic reduction (IMR) has been developed for rapid and on-site assay with very small volume of sample (i.e. less than 1ml whole blood). The reagent is a solution of homogeneously dispersed magnetic nanoparticles, which are coated with hydrophilic surfactants and bioprobes. Under external multiple alternating-current (ac) magnetic fields, magnetic nanoparticles oscillate with the multiple ac magnetic fields via magnetic interaction. The reagents under the external multiple ac magnetic fields show a magnetic property, called mixed-frequency ac magnetic susceptibility χac. Magnetic nanoparticles bind with the bioprobes on the outmost shell and become larger or clustered. The χac of the reagent is reduced, and the concentration of the biomolecules can be measured quantitatively. Several papers have demonstrated that IMR can be applied to assay proteins, viruses, chemicals, and nucleic acids once suitable bioprobes are immobilized onto the magnetic nanoparticles.

Rapid diagnosis of acute coronary syndrome (ACS) is a clinical and operational priority in busy emergency departments (ED). Since ACS is associated with a significant mortality and morbidity, early and correct diagnosis is of great importance. Chest pain is a frequent symptom in medical emergency departments and distinguishing patients with ACS within the chest pain group is a diagnostic challenge. Cardiac enzymes (including CPK/CK-MB, troponins, myoglobulin) and electrocardiography (ECG) in combination with the medical history and physical examination are at present the diagnostic cornerstones. Different cardiac enzymes are released after myocardial cell disintegration and are markers of cell necrosis, which might not be detected immediately after chest pain; and repeated measurements are suggested. Therefore novel biomarkers that rise earlier, have good diagnosis accuracy and have additional prognostic information are highly needed. Some publications address the potential benefit of the combination of multiple biomarker assays (markers of myocardial injury, inflammation/plaque ruptures or heart failure with different mechanism) could substantially increase clinical sensitivity and improve early risk stratification. However, this approach is rather time-consuming and not cost-effect. In the present study, a rapid IMR assay with multiple biomarkers is proposed and we will examine the performance of this new investigational IMR assays, comparison with current commercial assays.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with acute coronary syndrome

Exclusion Criteria: none

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute chest pain who are sent to the emergency departments will be included
Sampling Method: Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Diagnositic accuracy of acute myocardial infarction | 7 days
  Evaluation of the diagnostic performance of rapid IMR assays in detection of acute myocardial infarction; Cardiac enzymes (CPK/CK-MB, troponins), electrocardiography in combination with the symptoms of typical chest pain are at present the diagnostic gold standard.

SECONDARY OUTCOMES:
Combination of potential biomarkers in detection of ACS by rapid IMR system | 7 days
  Compared to cardiac enzymes (CK/CK-MB, troponin), the diagnostic performance of combination of new biomarkers (BNP, FABP4, CRP, etc.) in detection of ACS by rapid IMR system

OTHER OUTCOMES:
Prediction of MACEs by rapid IMR system | 6 months
  Evaluation of prognostic significance of multi-antibody-activated magnetic nanoparticles system (troponin, CK-MB, myoglobin, BNP, CRP, adipocyte fatty-acid binding protein/FABP-4) in acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, MD, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (3):
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District

IPD SHARING:
Plan to Share IPD: No